CLINICAL TRIAL: NCT06845527
Title: Characteristics and Outcomes of Outpatients Referred to an Gut Microbiota Clinic
Brief Title: Outcomes of Outpatients in an Gut Microbiota Clinic
Acronym: Microfec
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, IANIRO GIANLUCA, Principal Investigator, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: ID 6778
Record Dates: First submitted 2025-02-06; First posted 2025-02-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Intestinal Disease
Keywords: Gut Dysbiosis; Microbiome testing; Microbiome
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: The study cohort will consist of patients attending the Gut Microbiota Clinic at Policlinico Gemelli in Rome. Patients with all inclusion criteria and none of the exclusion criteria will be considered for this study. N=400 patients will be enrolled. Since the study is interventional and the primary objective is descriptive, the sample size justification is based on the precision of confidence intervals. This sample size will allow the calculation of 95% confidence intervals for the considered point estimates; these intervals will have a precision of at least 5% for categorical variables and a precision equal to one-tenth of the standard deviation for quantitative variables.
  Interventions: Other: Gut microbiome testing

INTERVENTIONS:
Other: Gut microbiome testing — Gut microbiome testing for the characterization of the patient gut microbiome

SUMMARY:
The gut microbiota plays a crucial role in human health, influencing metabolism, immunity, and pathogen resistance. Research has linked microbiome dysbiosis to various intestinal and extra-intestinal disorders, prompting interest in therapeutic strategies like fecal microbiota transplantation (FMT), which is now standard for recurrent Clostridioides difficile infection and shows promise for other conditions.

Despite its potential, the clinical integration of microbiome research remains limited due to biological complexity, lack of clinician awareness, and the absence of standardized guidelines. Meanwhile, patient demand for microbiome-based interventions is rising, leading some to seek non-scientific alternatives with potential health risks.

Since 2016, the Gut Microbiota Clinic at Fondazione Policlinico Gemelli has provided personalized microbiota-based treatments, collaborating with specialists across disciplines. The clinic primarily serves patients with gastrointestinal and extra-intestinal disorders and employs a multidisciplinary approach.

This study aims to characterize the clinical and microbiological profiles of patients attending the clinic and establish a microbiological database. Primary and secondary endpoints include microbiota composition changes and clinical outcomes assessed through validated diagnostic tools.

DETAILED DESCRIPTION:
The gut microbiota is a key mediator of various human functions, including metabolism, the immune system, and resistance to pathogen colonization. A growing body of scientific research has demonstrated-initially through association studies and subsequently through mechanistic experiments-that gut microbiome dysbiosis is linked to a wide range of both intestinal and extra-intestinal disorders.

This body of evidence has led to the exploration of gut microbiome modulation as a therapeutic strategy, such as fecal microbiota transplantation (FMT), which has become a standard treatment for recurrent Clostridioides difficile infection and has also shown promise for several other indications, including ulcerative colitis, irritable bowel syndrome, and metabolic syndrome.

Furthermore, there is increasing interest in leveraging the gut microbiome as a diagnostic tool in clinical practice for various applications, including disease diagnosis, prognosis, and risk assessment; prediction of patient response to specific therapies; guidance and personalization of microbiome-targeted interventions such as probiotics or FMT; and monitoring the effectiveness of these treatments.

Despite this enthusiasm, however, the integration of microbiome research advancements into routine clinical practice remains generally limited. This gap can be attributed to several factors, primarily the complexity of microbiome biology, the limited knowledge of gut microbiota among most healthcare professionals, and the absence of established guidelines and infrastructures for the clinical application of microbiome research.

In contrast to the relatively slow adoption of microbiome research by clinicians, there is growing enthusiasm and high expectations among various patient groups for the rapid implementation of microbiota-related findings in clinical practice. This discrepancy poses the risk of patients seeking alternative, non-scientific solutions due to the lack of medical guidance. As a result, many individuals turn to non-medical sources, often found online, which may expose them to potential health risks and significant financial costs.

Since 2016, the Gut Microbiota Clinic has been active within the CEMAD (Center for Digestive Diseases) at Fondazione Policlinico Gemelli. This clinic was established to address the needs of patients with gut microbiota imbalances, offering personalized therapeutic approaches based on microbiota profiling, which is assessed using a commercially available test. In particular, Fondazione Policlinico Gemelli collaborates with the company XBIOGEM for the production and supply of gut microbiota tests.

The clinic primarily evaluates patients with gastrointestinal disorders (e.g., irritable bowel syndrome, inflammatory bowel diseases, and colitis induced by oncological treatments) as well as other conditions (e.g. patients with autoimmune disorders or patients undergoing oncological treatments). It operates through close collaboration with specialists from other medical fields, depending on the patient's condition (e.g., gastroenterologists, rheumatologists, dermatologists, infectious disease specialists, etc.), and follows a multidisciplinary approach involving dietitians and psychologists/psychiatrists as needed.

This clinic is highly specialized and innovative and, to the best of our knowledge, is the first dedicated clinic of its kind worldwide.

The aim of our study is to describe the characteristics of patients attending the Gut Microbiota Clinic at Fondazione Policlinico Gemelli and to establish a clinical and microbiological database. This initiative seeks to bridge the gap between the vast diagnostic and therapeutic potential of the gut microbiome and its practical application in routine clinical care.

OBJECTIVES

Primary Objective The primary objective is to describe the clinical and microbiological characteristics of patients attending the Gut Microbiota Clinic at Fondazione Policlinico Gemelli.

Secondary Objectives

* To describe changes in microbiota composition in patients undergoing microbiota testing as part of routine clinical practice after receiving standard treatments.
* To assess clinical changes by evaluating follow-up consultations with the referring specialist (e.g., rheumatologist or dermatologist) for patients with extra-intestinal conditions, or through the judgment of the responsible physician. When applicable, validated diagnostic scores specific to the relevant condition (e.g., Mayo Score for ulcerative colitis, CDAI for Crohn's disease, or IBS-SSS for irritable bowel syndrome, PFS and OS for oncological patients) will be used.
* To establish a microbiological database.

ENDPOINTS

Primary Endpoint The primary endpoint is the assessment of the clinical and microbiological characteristics of patients attending the Gut Microbiota Clinic at Fondazione Policlinico Gemelli.

Secondary Endpoints

* Changes in microbiota composition in patients undergoing microbiota testing as part of routine clinical practice after receiving standard treatments.
* Clinical variations assessed by referring specialists using validated and disease-specific diagnostic scores.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Patient attending the Gut Microbiota Clinic at Fondazione Policlinico Universitario "A. Gemelli" IRCCS;
* Ability to provide informed consent for inclusion in the study;
* Patient in possession of a gut microbiota test, performed as part of routine clinical practice upon medical request, no more than one month prior to the first visit.

Exclusion Criteria:

* Age < 18 years;
* Severe psychiatric disorders;
* Inability to provide informed conse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients attending the Gut Microbiota Clinic at Fondazione Policlinico Universitario "A. Gemelli" IRCCS in possession of a gut microbiota test, performed as part of routine clinical practice upon medical request, no more than one month prior to the first visit.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-03-10 (Estimated); Study Completion 2027-03-10 (Estimated)

PRIMARY OUTCOMES:
Microbiological Characteristics of Patients at the Gut Microbiota Clinic | 24 months
  The microbiome test results that patients will bring to the visit will be analyzed, including:
  Alpha and beta diversity Taxonomic Composition (proportion of different bacterial phyla, genera, and species)

SECONDARY OUTCOMES:
Changes in Microbiota Composition in Patients Undergoing Routine Clinical Microbiota Testing After Standard Treatments | 24 months
  To describe changes in microbiota composition in patients undergoing microbiome testing as part of routine clinical practice after receiving standard treatments (Alpha and beta diversity, Taxonomic Composition - Proportion of different bacterial phyla, genera, and species).
Assessment of CDAI Scores | 24 months
  Crohn's Disease Activity Index (CDAI) for Crohn's disease (Range: 0-600; higher scores indicate worse disease activity)
Assessment of IBS-SSS | 24 months
  IBS Severity Scoring System (IBS-SSS) for irritable bowel syndrome (Range: 0-500; higher scores indicate worse symptoms).
Assessment of PFS Scores | 24 months
  Variation of of Progression-Free Survival (PFS) in cancers patients treated with immunotherapy or targeted therapies: In selected patients with a sustained response, PFS can exceed 24 to 48 months.
Pain intensity | 24 months
  The Visual Analog Scale (VAS) for Pain is a continuous scale, usually 10 cm long, where the patient marks the point that best represents their pain intensity. Scores range from 0 (no pain) to 10 (worst possible pain).
Assessment of OS scores | 24 months
  Description: Variation of Overall Survival (OS) in cancers patients treated with immunotherapy or targeted therapies: In selected patients with a sustained response, PFS can exceed 24 to 48 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
The individual data of patients will be shared
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Data will be given upon reasonable request to the PI

REFERENCES:
- [Background] Lin D, Medeiros DM. The microbiome as a major function of the gastrointestinal tract and its implication in micronutrient metabolism and chronic diseases. Nutr Res. 2023 Apr;112:30-45. doi: 10.1016/j.nutres.2023.02.007. Epub 2023 Mar 4. PMID 36965327
- [Background] Ghosh S, Whitley CS, Haribabu B, Jala VR. Regulation of Intestinal Barrier Function by Microbial Metabolites. Cell Mol Gastroenterol Hepatol. 2021;11(5):1463-1482. doi: 10.1016/j.jcmgh.2021.02.007. Epub 2021 Feb 18. PMID 33610769
- [Background] Zhang D, Jian YP, Zhang YN, Li Y, Gu LT, Sun HH, Liu MD, Zhou HL, Wang YS, Xu ZX. Short-chain fatty acids in diseases. Cell Commun Signal. 2023 Aug 18;21(1):212. doi: 10.1186/s12964-023-01219-9. PMID 37596634
- [Background] Horrocks V, King OG, Yip AYG, Marques IM, McDonald JAK. Role of the gut microbiota in nutrient competition and protection against intestinal pathogen colonization. Microbiology (Reading). 2023 Aug;169(8):001377. doi: 10.1099/mic.0.001377. PMID 37540126
- [Background] Martin AM, Sun EW, Rogers GB, Keating DJ. The Influence of the Gut Microbiome on Host Metabolism Through the Regulation of Gut Hormone Release. Front Physiol. 2019 Apr 16;10:428. doi: 10.3389/fphys.2019.00428. eCollection 2019. PMID 31057420
- [Background] Pedersen HK, Gudmundsdottir V, Nielsen HB, Hyotylainen T, Nielsen T, Jensen BA, Forslund K, Hildebrand F, Prifti E, Falony G, Le Chatelier E, Levenez F, Dore J, Mattila I, Plichta DR, Poho P, Hellgren LI, Arumugam M, Sunagawa S, Vieira-Silva S, Jorgensen T, Holm JB, Trost K; MetaHIT Consortium; Kristiansen K, Brix S, Raes J, Wang J, Hansen T, Bork P, Brunak S, Oresic M, Ehrlich SD, Pedersen O. Human gut microbes impact host serum metabolome and insulin sensitivity. Nature. 2016 Jul 21;535(7612):376-81. doi: 10.1038/nature18646. Epub 2016 Jul 13. PMID 27409811
- [Background] Pandey H, Jain D, Tang DWT, Wong SH, Lal D. Gut microbiota in pathophysiology, diagnosis, and therapeutics of inflammatory bowel disease. Intest Res. 2024 Jan;22(1):15-43. doi: 10.5217/ir.2023.00080. Epub 2023 Nov 8. PMID 37935653
- [Background] Yuan Y, Wang X, Huang S, Wang H, Shen G. Low-level inflammation, immunity, and brain-gut axis in IBS: unraveling the complex relationships. Gut Microbes. 2023 Dec;15(2):2263209. doi: 10.1080/19490976.2023.2263209. Epub 2023 Oct 2. PMID 37786296
- [Background] Moayyedi P, Surette MG, Kim PT, Libertucci J, Wolfe M, Onischi C, Armstrong D, Marshall JK, Kassam Z, Reinisch W, Lee CH. Fecal Microbiota Transplantation Induces Remission in Patients With Active Ulcerative Colitis in a Randomized Controlled Trial. Gastroenterology. 2015 Jul;149(1):102-109.e6. doi: 10.1053/j.gastro.2015.04.001. Epub 2015 Apr 7. PMID 25857665
- [Background] Rossen NG, Fuentes S, van der Spek MJ, Tijssen JG, Hartman JH, Duflou A, Lowenberg M, van den Brink GR, Mathus-Vliegen EM, de Vos WM, Zoetendal EG, D'Haens GR, Ponsioen CY. Findings From a Randomized Controlled Trial of Fecal Transplantation for Patients With Ulcerative Colitis. Gastroenterology. 2015 Jul;149(1):110-118.e4. doi: 10.1053/j.gastro.2015.03.045. Epub 2015 Mar 30. PMID 25836986
- [Background] Paramsothy S, Kamm MA, Kaakoush NO, Walsh AJ, van den Bogaerde J, Samuel D, Leong RWL, Connor S, Ng W, Paramsothy R, Xuan W, Lin E, Mitchell HM, Borody TJ. Multidonor intensive faecal microbiota transplantation for active ulcerative colitis: a randomised placebo-controlled trial. Lancet. 2017 Mar 25;389(10075):1218-1228. doi: 10.1016/S0140-6736(17)30182-4. Epub 2017 Feb 15. PMID 28214091
- [Background] El-Salhy M, Hatlebakk JG, Gilja OH, Brathen Kristoffersen A, Hausken T. Efficacy of faecal microbiota transplantation for patients with irritable bowel syndrome in a randomised, double-blind, placebo-controlled study. Gut. 2020 May;69(5):859-867. doi: 10.1136/gutjnl-2019-319630. Epub 2019 Dec 18. PMID 31852769